CLINICAL TRIAL: NCT07350759
Title: An Observational Study to Develop an Algorithm to Predict Decompensation of Congestive Heart Failure (dCHF) Using a Non-Invasive Wearable Device.
Brief Title: Observational Study Designed to Detect Decompensation of Congestive Heart Failure (dCHF) Using a Non-Invasive Wearable Device
Status: Not yet recruiting | Type: Observational
Sponsor: CHFDX,Inc. (Industry)
Collaborators: Tampa General Hospital (Other); University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY 008961
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Decompensated Chronic Heart Failure
Keywords: congestive heart failure; wearable monitor; predictive algrothim
MeSH Terms: conditions — Heart Failure | interventions — Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — saliva, plasma, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with congestive heart failure: Patients will be monitored by a a tiny, battery-free pressure sensor implanted in a branch of the pulmonary artery via a right-heart catheterization, previously placed for a history of decompensating heart failure.
  Interventions: Device: wearable ring device with multiple embedded sensors to detect heart rate, SVO2, respiratory rate, heart rate variability and a number of other related physiologic parameters

INTERVENTIONS:
Device: wearable ring device with multiple embedded sensors to detect heart rate, SVO2, respiratory rate, heart rate variability and a number of other related physiologic parameters — In this observational study, a non-invasive, wearable ring used for continuous passive collection of physiologic data (sleep, activity, heart rate, HRV, temperature) will be used to collect data from all patients in the study. Data are used solely for research and algorithm development and are not used for diagnosis or treatment.

SUMMARY:
This is a prospective, observational pilot study designed to develop a mathematical algorithm capable of predicting decompensation of congestive heart failure (dCHF) using physiologic data collected from a non-invasive wearable device. Participants with a remote hemodynamic pulmonary artery pressure monitor will wear a wearable device continuously for up to 12 months. Wearable data will be analyzed in relation to the hemodynamic monitor defined sentinel events of heart failure decompensation to identify predictive signal patterns. Optional biospecimen (DNA, blood, urine) and voice sample collection will support future biomarker discovery.

DETAILED DESCRIPTION:
Participants with chronic congestive heart failure and using a pulmonary artery pressure monitor will be enrolled and followed for a minimum of 6 months and up to 12 months. Daily pulmonary artery (PA) pressures obtained via the remote monitoring device will serve as the reference standard for identifying decompensated CHF events ("sentinel events"), defined by sustained elevations in PA diastolic pressure associated with medication changes by the clinical care team.

Physiologic data from the wearable-including heart rate, heart rate variability, sleep metrics, activity levels, oxygen saturation and temperature-will be collected continuously and analyzed in the 1-7 days preceding and following sentinel events. Time-series statistical methods and machine-learning models will be used to develop a predictive algorithm for dCHF.

Participants may opt in to optional biospecimen collection (cheek swab DNA, plasma, urine) and weekly voice recordings to support future research into biomarkers and digital phenotypes associated with heart failure decompensation. The wearable data are not used for clinical decision-making, and all participants continue to receive standard heart failure care.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years

  * Current use of a hemodynamic sensoring device
  * At least 4 consecutive weeks of stabilized "goal" pulmonary artery pressures
  * Access to a personal smartphone with Wi-Fi or cellular connectivity

Exclusion Criteria:

* • Inability to provide informed consent

  * Inability to read or understand English
  * Likely non-adherence to wearable device use
  * Prisoners
  * Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of South Florida Tampa General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in multiple physiologic parameters from baseline that correlate with onset of dCHF | Up to 12 Months
  Identification of reproducible changes in wearable physiologic data that occur in the 1-7 days preceding a hemodynamic monitoring device detection of elevated pulmonary artery pressure sustained over 2 days defined as a sentinel event of decompensated CHF.

CONTACTS AND LOCATIONS:
Overall Officials: Wu, DO, Principal Investigator — Tampa General Hospital
Locations (2):
- United States (2):
  - USF Office of Clinical Research, Tampa, Florida
  - USF, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
Observational data only being collected to produce a predictive algorithm IPD is not required for this goal.

REFERENCES:
- [Background] Shavelle DM, Desai AS, Abraham WT, Bourge RC, Raval N, Rathman LD, Heywood JT, Jermyn RA, Pelzel J, Jonsson OT, Costanzo MR, Henderson JD, Brett ME, Adamson PB, Stevenson LW; CardioMEMS Post-Approval Study Investigators. Lower Rates of Heart Failure and All-Cause Hospitalizations During Pulmonary Artery Pressure-Guided Therapy for Ambulatory Heart Failure: One-Year Outcomes From the CardioMEMS Post-Approval Study. Circ Heart Fail. 2020 Aug;13(8):e006863. doi: 10.1161/CIRCHEARTFAILURE.119.006863. Epub 2020 Aug 6. PMID 32757642
- [Background] Abraham WT, Adamson PB, Bourge RC, Aaron MF, Costanzo MR, Stevenson LW, Strickland W, Neelagaru S, Raval N, Krueger S, Weiner S, Shavelle D, Jeffries B, Yadav JS; CHAMPION Trial Study Group. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomised controlled trial. Lancet. 2011 Feb 19;377(9766):658-66. doi: 10.1016/S0140-6736(11)60101-3. PMID 21315441
- [Background] Desai AS, Bhimaraj A, Bharmi R, Jermyn R, Bhatt K, Shavelle D, Redfield MM, Hull R, Pelzel J, Davis K, Dalal N, Adamson PB, Heywood JT. Ambulatory Hemodynamic Monitoring Reduces Heart Failure Hospitalizations in "Real-World" Clinical Practice. J Am Coll Cardiol. 2017 May 16;69(19):2357-2365. doi: 10.1016/j.jacc.2017.03.009. Epub 2017 Mar 19. PMID 28330751
- [Background] 8. JoAnn Lindenfeld, on behalf of the GUIDE-HF, CHAMPION, and LAPTOPHF investigators. Longer Term Effects of Hemodynamic Monitoring on Outcomes: A Combined Data Analysis of patients with HFrEF in CHAMPION, GUIDE-HF, and LAPTOP-HF. Presented at THT Conference, Boston, MA, March 2023.
- [Background] Abraham WT, Stevenson LW, Bourge RC, Lindenfeld JA, Bauman JG, Adamson PB; CHAMPION Trial Study Group. Sustained efficacy of pulmonary artery pressure to guide adjustment of chronic heart failure therapy: complete follow-up results from the CHAMPION randomised trial. Lancet. 2016 Jan 30;387(10017):453-61. doi: 10.1016/S0140-6736(15)00723-0. Epub 2015 Nov 9. PMID 26560249
- [Background] Givertz MM, Stevenson LW, Costanzo MR, Bourge RC, Bauman JG, Ginn G, Abraham WT; CHAMPION Trial Investigators. Pulmonary Artery Pressure-Guided Management of Patients With Heart Failure and Reduced Ejection Fraction. J Am Coll Cardiol. 2017 Oct 10;70(15):1875-1886. doi: 10.1016/j.jacc.2017.08.010. PMID 28982501
- [Background] Adamson PB. Pathophysiology of the transition from chronic compensated and acute decompensated heart failure: new insights from continuous monitoring devices. Curr Heart Fail Rep. 2009 Dec;6(4):287-92. doi: 10.1007/s11897-009-0039-z. PMID 19948098
- [Background] Redfield MM. Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2016 Nov 10;375(19):1868-1877. doi: 10.1056/NEJMcp1511175. No abstract available. PMID 27959663
- [Background] Ellison DH, Felker GM. Diuretic Treatment in Heart Failure. N Engl J Med. 2017 Nov 16;377(20):1964-1975. doi: 10.1056/NEJMra1703100. No abstract available. PMID 29141174
- [Background] Scott MC, Winters ME. Congestive Heart Failure. Emerg Med Clin North Am. 2015 Aug;33(3):553-62. doi: 10.1016/j.emc.2015.04.006. Epub 2015 Jun 10. PMID 26226866
- [Background] Chen J, Aronowitz P. Congestive Heart Failure. Med Clin North Am. 2022 May;106(3):447-458. doi: 10.1016/j.mcna.2021.12.002. Epub 2022 Apr 4. PMID 35491065